CLINICAL TRIAL: NCT01052480
Title: A Randomized, Open-Label, Phase 2, Multicenter Safety and Exploratory Efficacy Study of Investigational Anti-Influenza Immune Plasma for the Treatment of Influenza (IRC002)
Brief Title: Safety and Efficacy of Investigational Anti-Influenza Immune Plasma in Treating Influenza
Acronym: IRC002
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-I-0043; IRC002 (Other: NIAID Influenza Research Collaboration)
Record Dates: First submitted 2010-01-16; First posted 2010-01-20 (Estimated); Results first posted 2017-05-23 (Actual); Last update posted 2017-09-05 (Actual); Status verified 2017-06

CONDITIONS: Influenza A; Influenza B
Keywords: Antiviral; Anti-Influenza Immune Plasma; Emerging Infectious Disease; Swine Flu
MeSH Terms: conditions — Communicable Diseases, Emerging; Orthomyxoviridae Infections | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Plasma and Standard Care (Experimental): Participants will receive plasma with high titer anti-influenza A or anti-influenza B antibodies (Anti-Influenza Immune Plasma) in addition to standard care.
  Interventions: Biological: Anti-Influenza Immune Plasma; Drug: Standard Care
- Standard Care (Active Comparator): Participants will receive standard care.
  Interventions: Drug: Standard Care

INTERVENTIONS:
Biological: Anti-Influenza Immune Plasma — 2 units of plasma with high titer anti-influenza A or anti-influenza B antibodies at baseline
  Arms: Plasma and Standard Care
Drug: Standard Care — All subjects will receive an anti-influenza antiviral (e.g., oseltamivir or zanamivir), but may include treatment with licensed antivirals in patient populations or at doses not covered in the package insert, or with medications available under a EUA. Standard care may also include antibiotics and other medications.

SUMMARY:
This randomized, open-label, multicenter phase 2 trial will assess the safety, efficacy, and pharmacokinetics (PK) of anti-influenza plasma in subjects with influenza A or B. Hospitalized subjects with influenza A or B that have either a low oxygen level or a high respiratory rate will be eligible for study participation. This study will enroll adults, children and pregnant women.

DETAILED DESCRIPTION:
Morbidity and mortality occur despite treatment with current antivirals. Circulating influenza H1N1 and H3N2 isolates are highly resistant to amantadine and rimantadine, whereas previous seasonal H1N1 isolates were highly resistant to oseltamivir. So there is concern that circulating influenza A/H1N1 2009 virus may also acquire oseltamivir resistance.

This randomized, open-label, multicenter phase 2 trial will assess the safety, efficacy, and pharmacokinetics (PK) of anti-influenza plasma in subjects with influenza. Hospitalized subjects with influenza at risk for severe disease (as defined in the inclusion criteria) will be eligible for study participation. This study will enroll adults, children and pregnant women.

Up to 40 sites in the United States will participate in this protocol. One hundred eligible subjects will be randomized in a 1:1 ratio to receive either 2 units (or pediatric equivalent) of anti-influenza immune plasma on Study Day 0 in addition to standard care or standard care alone (50 subjects receiving standard care alone; 50 subjects receiving anti-influenza immune plasma and standard care).

Subjects will be assessed on Study Day 0 (pre-dose), 30 minutes post-dose (plasma arm only), and on Study Days 1, 2, 4, 7, 14, and 28. All subjects will undergo a series of efficacy, safety, and PK (HAI) assessments during the study. Blood samples will be collected at each time point (except Day 1). Nasal and oropharyngeal swabs for influenza PCR will be obtained on Days 0,1,2,4 and 7.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of influenza A or B within 72 hours prior to enrollment (by local assay including rapid antigen, direct fluorescent antibody (DFA), polymerase chain reaction (PCR), or culture, and must be able to detect and distinguish influenza A from influenza B)
* Hospitalization for signs and symptoms of influenza (decision for hospitalization will be up to the individual treating clinician).
* Abnormal respiratory status, defined as room air saturation of oxygen (SaO2) less than 93% or tachypnea (respiratory rate above an age adjusted normal range)
* Agree to the storage of specimens and data
* ABO compatible plasma available on site or available within 24 hours after randomization with activity against locally circulating strains of influenza

Exclusion Criteria:

* Receipt of non-licensed treatment for influenza within the last 2 weeks (or plans to receive any time during the study). This does not include licensed drugs at non approved doses, off-label indications, or drugs available under an Emergency Use Authorization (EUA).
* History of severe allergic reaction to blood products (as judged by the investigator).
* Medical conditions for which receipt of 500 mL volume (or 8 mL/kg for pediatric patients) may be dangerous to the subject (e.g. decompensated congestive heart failure [CHF], etc.)
* Clinical suspicion that etiology of acute illness is primarily due to a condition other than active influenza virus replication (e.g., a bacterial or fungal infection)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Beigel, MD, Study Chair — Leidos Biomedical Research, Inc. in support of Laboratory of Immunoregulation, NIAID, NIH; Richard Davey, MD, Study Chair — Laboratory of Immunoregulation, NIAID, NIH
Locations (35):
- United States (35):
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - Naval Medical Center San Diego, San Diego, California
  - Los Angeles Biomedical Research Institute, CA, Torrance, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Washington, DC VA Med Center, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Northwestern University (NU), Chicago, Illinois
  - The Rush University Medical Center, Chicago, Illinois
  - University of Maryland School of Medicine Center for Vaccine Development, Baltimore, Maryland
  - John Hopkins University (JHU), Baltimore, Maryland
  - Walter Reed National Military Medical Center (WRNMMC), Bethesda, Maryland
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital/Harvard Medical School, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston Med Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Bronson Healthcare Group, Kalamazoo, Michigan
  - Saint Mary's Hospital (Mayo Clinic), Rochester, Minnesota
  - Mount Sinai Medical Center, New York, New York
  - Cornell Clinical Trials Unit, New York Presbyterian Hospital, Weill Cornell Medical College, New York, New York
  - Montefiore Medical Center/Albert Einstein College of Medicine, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - University of Cincinnati College of Medicine, Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center (UPMC), Pittsburgh, Pennsylvania
  - Texas Tech University Health Science Center (HSC)- Amarillo, Amarillo, Texas
  - Texas Children's Hospital, Houston, Texas
  - Texas Tech HSC-Lubbock, TX, Lubbock, Texas
  - Naval Medical Center Portsmouth, Portsmouth, Virginia
  - Madigan Army Medical Center (MAMC), Tacoma, Washington

REFERENCES:
- [Background] Morse SS. Factors in the emergence of infectious diseases. Emerg Infect Dis. 1995 Jan-Mar;1(1):7-15. doi: 10.3201/eid0101.950102. PMID 8903148
- [Background] Bean WJ, Schell M, Katz J, Kawaoka Y, Naeve C, Gorman O, Webster RG. Evolution of the H3 influenza virus hemagglutinin from human and nonhuman hosts. J Virol. 1992 Feb;66(2):1129-38. doi: 10.1128/JVI.66.2.1129-1138.1992. PMID 1731092
- [Background] de Jong MD, Tran TT, Truong HK, Vo MH, Smith GJ, Nguyen VC, Bach VC, Phan TQ, Do QH, Guan Y, Peiris JS, Tran TH, Farrar J. Oseltamivir resistance during treatment of influenza A (H5N1) infection. N Engl J Med. 2005 Dec 22;353(25):2667-72. doi: 10.1056/NEJMoa054512. PMID 16371632
- [Derived] Beigel JH, Tebas P, Elie-Turenne MC, Bajwa E, Bell TE, Cairns CB, Shoham S, Deville JG, Feucht E, Feinberg J, Luke T, Raviprakash K, Danko J, O'Neil D, Metcalf JA, King K, Burgess TH, Aga E, Lane HC, Hughes MD, Davey RT; IRC002 Study Team. Immune plasma for the treatment of severe influenza: an open-label, multicentre, phase 2 randomised study. Lancet Respir Med. 2017 Jun;5(6):500-511. doi: 10.1016/S2213-2600(17)30174-1. Epub 2017 May 15. PMID 28522352
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/detail/B_2010-I-0043.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Plasma and Standard Care: Participants will receive plasma with high titer anti-influenza A or anti-influenza B antibodies in addition to standard care.
  Anti-Influenza Immune Plasma: 2 units of plasma with high titer anti-influenza A or anti-influenza B antibodies at baseline
  Standard Care: Standard care for hospitalized people with influenza
- Standard Care: Participants will receive standard care.
  Standard Care: Standard care for hospitalized people with influenza
Period: Overall Study
Arm/Group | Plasma and Standard Care | Standard Care
Started | 49 | 49
Completed | 41 | 32
Not Completed | 8 | 17
Not completed — Lost to Follow-up | 3 | 3
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 3 | 7
Not completed — Physician Decision | 0 | 2
Not completed — Death | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Plasma and Standard Care | Standard Care | Total
Number analyzed (Participants) | 49 | 49 | 98
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 50 [38 to 66] | 57 [39 to 71] | 53 [38 to 69]
Age, Customized [Count of Participants; unit: Participants] — The <18 and >=18 categories match a protocol-specified division, so it is most appropriate to present categorized age this way.
  Participants
    <18 | 4 | 7 | 11
    >=18 | 45 | 42 | 87
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 27 | 51
  Male | 25 | 22 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 6 | 10
  Not Hispanic or Latino | 43 | 39 | 82
  Unknown or Not Reported | 2 | 4 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 16 | 9 | 25
  White | 29 | 32 | 61
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Time to Normalization of Respiratory Status (Primary Efficacy Population)
Description: Normalized respiratory status is defined as room air saturation of oxygen [SaO2] greater than or equal to 93% AND respiratory rate within normal ranges.
Time Frame: Measured from Day 0 through Day 28
Population: The population analyzed is the Primary Efficacy Population (PEP), defined as the subset of randomized participants who tested positive for influenza.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Plasma and Standard Care | Standard Care
Number analyzed (Participants) | 42 | 45
days | 7 [2 to NA] — Upper quartile is not available because fewer than 75% of the analyzed participants achieved normalized respiratory status. Lower quartile and median were estimated from Kaplan-Meier analysis. | 28 [7 to NA] — Upper quartile is not available because fewer than 75% of the analyzed participants achieved normalized respiratory status. Lower quartile and median were estimated from Kaplan-Meier analysis.
Statistical Analysis 1: Comparison: Plasma and Standard Care vs Standard Care; Test type: Superiority or Other; p = 0.069, Log Rank

2. Secondary Outcome: Time to Normalization of Respiratory Status (All Randomized Participants)
Description: as for outcome 1
Time Frame: Measured from Day 0 through Day 28
Population: All randomized participants
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Plasma and Standard Care | Standard Care
Number analyzed (Participants) | 49 | 49
days | 14 [2 to NA] — Upper quartile is not available because fewer than 75% of the analyzed participants achieved normalized respiratory status. Lower quartile and median were estimated from Kaplan-Meier analysis. | NA [7 to NA] — Median and upper quartile are not available because fewer than 50% of the analyzed participants achieved normalized respiratory status. Lower quartile was estimated from Kaplan-Meier analysis.

3. Secondary Outcome: Duration of Time to Resolution of Clinical Symptoms
Description: The assessed clinical symptoms were nausea, vomiting, diarrhea, sore throat, headache, muscle ache, cough, and shortness of breath. Symptoms were assessed at days 0, 1, 2, 4, 7, 14, and 28.
Time Frame: Measured from Day 0 through Day 28
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Plasma and Standard Care | Standard Care
Number analyzed (Participants) | 42 | 45
days | NA [14 to NA] — Median and upper quartile are not available because fewer than 50% of the analyzed participants had symptoms resolved. Lower quartile was estimated from Kaplan-Meier analysis | NA [28 to NA] — Median and upper quartile are not available because fewer than 50% of the analyzed participants had symptoms resolved. Lower quartile was estimated from Kaplan-Meier analysis

4. Secondary Outcome: Duration of Time to Resolution of Fever
Description: Fever was defined as either a temperature > 38.0 C, or a report of a Grade 1 or higher fever as an adverse event.
Time Frame: Measured from Day 0 through Day 28
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Plasma and Standard Care | Standard Care
Number analyzed (Participants) | 42 | 45
days | NA [0 to NA] — Median and upper quartile are not available because nearly all participants had no fever at Day 0. Lower quartile was estimated from Kaplan-Meier analysis. | NA [0 to NA] — Median and upper quartile are not available because nearly all participants had no fever at Day 0. Lower quartile was estimated from Kaplan-Meier analysis.

5. Secondary Outcome: Duration of Time to Resolution of All Symptoms and Fever
Description: The assessed symptoms were nausea, vomiting, diarrhea, sore throat, headache, muscle ache, cough, and shortness of breath. Fever was defined as either a temperature > 38.0 C, or a report of a Grade 1 or higher fever as an adverse event.
Time Frame: Measured from Day 0 through Day 28
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Plasma and Standard Care | Standard Care
Number analyzed (Participants) | 42 | 45
days | NA [14 to NA] — Median and upper quartile are not available because fewer than 50% of the analyzed participants had all symptoms and fever resolved. Lower quartile was estimated from Kaplan-Meier analysis. | NA [28 to NA] — Median and upper quartile are not available because fewer than 50% of the analyzed participants had all symptoms and fever resolved. Lower quartile was estimated from Kaplan-Meier analysis.

6. Secondary Outcome: Time to 20% Improvement in Sequential Organ Failure Assessment (SOFA) Score for Participants >= 18 Years Old and Pediatric Logistic Organ Dysfunction (PELOD) Score for Participants < 18 Years Old
Description: The analysis is restricted to participants >= 18 years old and the SOFA score because there were very few evaluations of the PELOD score during follow-up for the participants < 18 years old. The adult population was further subset to those with a non-missing and non-zero SOFA score at Day 0; those with missing SOFA score at Day 0 did not have a starting point, and those with SOFA = 0 at Day 0 could not have an improvement.
Time Frame: Measured from Day 0 through Day 28
Population: The population analyzed is the Primary Efficacy Population (PEP), defined as the subset of randomized participants who tested positive for influenza. This subset was further restricted to those >= 18 years with an available (non-zero) Day 0 SOFA evaluation.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Plasma and Standard Care | Standard Care
Number analyzed (Participants) | 28 | 33
days | 4 [2 to NA] — Upper quartile is not available because fewer than 75% of the analyzed participants had 20% improvement in SOFA score. Median and lower quartile were estimated from Kaplan-Meier analysis. | 28 [7 to NA] — Upper quartile is not available because fewer than 75% of the analyzed participants had 20% improvement in SOFA score. Median and lower quartile were estimated from Kaplan-Meier analysis.

7. Secondary Outcome: 50 Millimeters of Mercury (mm/Hg) Improvement in PaO2/FiO2 Ratio Over Time
Description: Number of participants with ABG done and no increase of 50 millimeters of mercury (mm/Hg) or greater in PaO2/FiO2 ratio. PaO2/FiO2 ratio was evaluated by an ABG. ABG was performed only when clinically indicated.
Time Frame: Measured at Days 1, 2, 4, 7, 14, 28
Population: The population analyzed is the Primary Efficacy Population (PEP), defined as the subset of randomized participants who tested positive for influenza. This subset was further restricted to those participants with a PaO2/FiO2 ratio (ABG performed) at Day 0.
Measure: Number; unit: participants
Arm/Group | Plasma and Standard Care | Standard Care
Number analyzed (Participants) | 25 | 29
participants
  Day 1 | 11 | 14
  Day 2 | 12 | 12
  Day 4 | 7 | 11
  Day 7 | 7 | 9
  Day 14 | 3 | 5
  Day 28 | 2 | 3

8. Secondary Outcome: In-hospital Mortality
Description: Number of deaths in hospital during initial hospital admission
Time Frame: Measured from Day 0 through Day 28
Population: All randomized participants
Measure: Number; unit: participants
Arm/Group | Plasma and Standard Care | Standard Care
Number analyzed (Participants) | 49 | 49
participants | 1 | 5

9. Secondary Outcome: 28-day Mortality
Description: Number of deaths during study follow-up
Time Frame: Measured from Day 0 through Day 28
Population: All randomized participants
Measure: Number; unit: participants
Arm/Group | Plasma and Standard Care | Standard Care
Number analyzed (Participants) | 49 | 49
participants | 1 | 5

10. Secondary Outcome: Duration of Hospitalization
Description: Days that a participant spent at the hospital. Multiple hospitalizations are summed up.
Time Frame: Measured from Day 0 through Day 28
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Plasma and Standard Care | Standard Care
Number analyzed (Participants) | 42 | 45
days | 6 [4 to 16] | 11 [5 to 25]

11. Secondary Outcome: Number of ICU Admissions
Description: Number of ICU admissions during study follow-up. The intent was to analyze any number of ICU admissions.
Time Frame: Measured from Day 0 through Day 28
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Plasma and Standard Care | Standard Care
Number analyzed (Participants) | 42 | 45
participants
  1 ICU admission | 40 | 38
  2 ICU admissions | 2 | 5
  4 ICU admissions | 0 | 2

12. Secondary Outcome: Duration of Stay in ICU
Description: Days that a participant spent in ICU. Multiple ICU admissions are summed up.
Time Frame: Measured from Day 0 through Day 28
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Plasma and Standard Care | Standard Care
Number analyzed (Participants) | 42 | 45
days | 2.5 [0 to 9] | 3 [0 to 13]

13. Secondary Outcome: Days on Supplemental Oxygen
Description: Time (in days) of supplemental oxygen use
Time Frame: Measured from Day 0 through Day 28
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Plasma and Standard Care | Standard Care
Number analyzed (Participants) | 42 | 45
days | 7 [1 to 28] | 8 [3 to 28]

14. Secondary Outcome: Duration of Supplemental Oxygen
Description: Duration of supplemental oxygen use in days
Time Frame: Measured from Day 0 through Day 28
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Plasma and Standard Care | Standard Care
Number analyzed (Participants) | 42 | 45
days | 7 [1 to 28] | 8 [3 to 28]

15. Secondary Outcome: Incidence of Acute Respiratory Distress Syndrome (ARDS) Present
Description: Incidence of participants with acute respiratory distress syndrome (ARDS), restricted to those without ARDS at Day 0.
Time Frame: Measured at Days 0, 1, 2, 4, 7, 14, 28
Population: The population analyzed is the Primary Efficacy Population (PEP), defined as the subset of randomized participants who tested positive for influenza. This population is further restricted to those participants who did not have ARDS at Day 0.
Measure: Number; unit: participants
Arm/Group | Plasma and Standard Care | Standard Care
Number analyzed (Participants) | 28 | 26
participants | 0 | 3

16. Secondary Outcome: Days on Mechanical Ventilation
Description: Time (in days) of mechanical ventilation use
Time Frame: Measured from Day 0 through Day 28
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Plasma and Standard Care | Standard Care
Number analyzed (Participants) | 42 | 45
days | 0 [0 to 6] | 3 [0 to 14]

17. Secondary Outcome: Duration of Mechanical Ventilation
Description: Duration of mechanical ventilation use in days. Multiple mechanical ventilation durations are summed up.
Time Frame: Measured from Day 0 through Day 28
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Plasma and Standard Care | Standard Care
Number analyzed (Participants) | 42 | 45
days | 0 [0 to 6] | 3 [0 to 14]

18. Secondary Outcome: Disposition Following Initial Hospitalization
Description: Disposition following initial hospitalization was categorized as follows: "released home - home health care not required", " released home with home health care", "transferred to long-term care facility", "hospitalization ongoing at Day 28", "deceased".
Time Frame: Measured from Day 0 through Day 28
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Plasma and Standard Care | Standard Care
Number analyzed (Participants) | 42 | 45
participants
  released home - home health care not required | 21 | 17
  released home with home health care | 9 | 6
  transferred to long-term care facility | 4 | 6
  hospitalization ongoing at Day 28 | 7 | 9
  deceased | 1 | 5

19. Secondary Outcome: Duration of Viral Shedding < Lower Limit of Quantification (LLOQ) in Nasal Swabs
Description: Duration of viral shedding < lower limit of quantification (LLOQ) in nasal swabs (restricted to participants with viral shedding >= LLOQ in nasal swabs at Day 0)
Time Frame: Measured from Day 0 through Day 28
Population: The population analyzed is the Primary Efficacy Population (PEP), defined as the subset of randomized participants who tested positive for influenza. This subset was further restricted to those participants with viral shedding >= LLOQ in nasal swabs at Day 0.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Plasma and Standard Care | Standard Care
Number analyzed (Participants) | 27 | 35
days | 1 [1 to NA] — Upper quartile is not available because fewer than 75% of the analyzed participants had viral shedding < LLOQ in nasal swabs. Lower quartile and median were estimated from Kaplan-Meier analysis. | 1 [1 to NA] — Upper quartile is not available because fewer than 75% of the analyzed participants had viral shedding < LLOQ in nasal swabs. Lower quartile and median were estimated from Kaplan-Meier analysis.

20. Secondary Outcome: Incidence and Week of Gestation of Delivery of a Live Pre-term Infant for Pregnant Women
Description: Incidence and week of gestation of delivery of a live pre-term infant for pregnant female participants
Time Frame: Measured through to Day 28
Population: Measure was not analyzed since there was only one pregnant participant. No aggregate results were available for posting, and the individual participant-level data were not posted due to being potentially identifiable.
Arm/Group | Plasma and Standard Care | Standard Care
Number analyzed (Participants) | 0 | 0

21. Secondary Outcome: Incidence and Duration of Pre-term Labor (Defined as Labor Occurring < 36 Weeks) for Pregnant Women
Description: Incidence and duration of pre-term labor (defined as labor occurring < 36 weeks) for pregnant female participants
Time Frame: Measured through Day 28
Population: as for outcome 20
Arm/Group | Plasma and Standard Care | Standard Care
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Incidence of Spontaneous Abortion or Stillborn Fetus for Pregnant Women
Description: Incidence of spontaneous abortion or stillborn fetus for pregnant female participants
Time Frame: Measured from Day 0 through Day 28
Population: as for outcome 20
Arm/Group | Plasma and Standard Care | Standard Care
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the conduct of the study; from Day 0 to Day 28
Description: Adverse events were assessed by treatment received (as opposed to randomized treatment).The Participant Flow is presented by randomized treatment.
Arm/Group | Plasma and Standard Care | Standard Care
All-Cause Mortality (participants affected / at risk) | 1/49 | 5/49
Serious Adverse Events (participants affected / at risk) | 9/46 | 20/52
Other Adverse Events (participants affected / at risk) | 36/46 | 29/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Plasma and Standard Care (N=46) | Standard Care (N=52)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 2
Cerebral infarction (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 0 | 1
Sedation (Nervous system disorders) | 0 | 1
Mental impairment (Nervous system disorders) | 0 | 1
Septic shock (Infections and infestations) | 1 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Lower respiratory tract infection viral (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Abdominal compartment syndrome (Gastrointestinal disorders) | 0 | 1
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 2
Gout (Metabolism and nutrition disorders) | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Hepatic haematoma (Hepatobiliary disorders) | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1
Liver injury (Hepatobiliary disorders) | 1 | 0
Blood creatine phosphokinase MB increased (Investigations) | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Endotracheal intubation (Surgical and medical procedures) | 0 | 2
Thoracostomy (Surgical and medical procedures) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Shock (Vascular disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Plasma and Standard Care (N=46) | Standard Care (N=52)
Blood glucose increased (Investigations) | 5 | 6
Aspartate aminotransferase increased (Investigations) | 5 | 5
Blood albumin decreased (Investigations) | 4 | 4
Blood creatinine increased (Investigations) | 3 | 3
Blood uric acid increased (Investigations) | 1 | 4
Alanine aminotransferase increased (Investigations) | 1 | 4
Blood sodium decreased (Investigations) | 3 | 2
Haemoglobin decreased (Investigations) | 2 | 3
Blood bilirubin increased (Investigations) | 1 | 3
Blood sodium increased (Investigations) | 1 | 3
Blood creatine phosphokinase increased (Investigations) | 3 | 1
Lymphocyte count decreased (Investigations) | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 5 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 2
Alkalosis (Metabolism and nutrition disorders) | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 8 | 2
Nausea (Gastrointestinal disorders) | 6 | 2
Vomiting (Gastrointestinal disorders) | 0 | 3
Constipation (Gastrointestinal disorders) | 3 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 5
Anaemia (Blood and lymphatic system disorders) | 5 | 4
Leukopenia (Blood and lymphatic system disorders) | 3 | 1
Pyrexia (General disorders) | 5 | 5
Headache (Nervous system disorders) | 5 | 2
Hypotension (Vascular disorders) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No